CLINICAL TRIAL: NCT06386861
Title: Developing Culturally-Tailored Interventions to Overcome Genomic Health Disparities in Communities of Color
Brief Title: Validating the Spanish "Attitudes Toward Genomics and Precision Medicine" (AGPM).
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24.210.01e
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Adult ALL
Keywords: genomics; precision medicine; attitudes and beliefs; health literacy; health numeracy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Behavior | interventions — Precision Medicine

STUDY DESIGN:
Intervention Model Description: 500 English-speaking individuals identifying as Hispanic, Latino, or Latina 500 Spanish-speaking individuals identifying as Hispanic, Latino, or Latina
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGPM for English Speakers (Other): Participants identifying as Hispanic, Latino, or Latina whose primary language is English
  Interventions: Other: Attitudes Toward Genomics and Precision Medicine (English)
- AGPM for Spanish Speakers (Other): Participants identifying as Hispanic, Latino, or Latina whose primary language is Spanish
  Interventions: Other: Attitudes Toward Genomics and Precision Medicine (Spanish)

INTERVENTIONS:
Other: Attitudes Toward Genomics and Precision Medicine (English) — completing the English version of the AGPM and validated health literacy and numeracy instruments
  Arms: AGPM for English Speakers
Other: Attitudes Toward Genomics and Precision Medicine (Spanish) — completing the Spanish version of the AGPM and validated health literacy and numeracy instruments
  Arms: AGPM for Spanish Speakers

SUMMARY:
The investigators aim to evaluate English and Spanish versions of the "Attitudes toward genomics and precision medicine" instrument (AGPM). This study will help validating a Spanish version of the AGPM among people identifying as Hispanic, Latino, or Latina. Having a valid instrument is important for developing tailored interventions to decrease disparities in genomic healthcare for this population.

DETAILED DESCRIPTION:
The investigators will recruit 1,000 individuals (500 English-speaking and 500 Spanish-speaking) to complete the AGPM and previously validated instruments assessing health literacy and numeracy. Results will establish the psychometric properties of the Spanish version of the AGPM.

ELIGIBILITY:
Inclusion Criteria:

* adult (18+ yrs.)
* identifying as Hispanic, Latino, or Latina
* able to provide opt-in electronic informed consent

Exclusion Criteria:

* under age 18 yrs.
* not identifying as Hispanic, Latino, or Latina
* not able to provide opt-in electronic informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychometric properties | up to two weeks
  Establish the psychometric properties of the translated AGPM

SECONDARY OUTCOMES:
Health literacy/numeracy | up to two weeks
  Establish correlations between health literacy/numeracy and AGPM scores

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Dwyer, PhD, Principal Investigator — Boston College
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the developers of the AGPM
Supporting Information: ICF
Time Frame: Following publication, available indefinitely through the developers of the AGPM
Access Criteria: Must contact the AGPM developers

REFERENCES:
- [Background] DuBois JM, Mozersky J, Antes A, English T, Parsons MV, Baldwin K. Attitudes toward genomics and precision medicine. J Clin Transl Sci. 2021 Apr 8;5(1):e120. doi: 10.1017/cts.2021.774. eCollection 2021. PMID 34267947